CLINICAL TRIAL: NCT02812342
Title: Topical Tofacitinib for the Treatment of Alopecia Areata and Its Variants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1510016586
Record Dates: First submitted 2016-06-21; First posted 2016-06-24 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Alopecia Areata; Alopecia Totalis; Alopecia Universalis
Keywords: Alopecia
MeSH Terms: conditions — Alopecia Areata; Alopecia universalis; Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tofacitinib ointment (Experimental): Patients with AA (with at least 2 patches of alopecia involving the scalp), AT or AU will be treated with tofacitinib ointment for a maximum of 6 months. During treatment, patients will be evaluated every 4 weeks and effectiveness of the medication will be measured by changes in hair growth.
  Interventions: Drug: Tofacitinib ointment

INTERVENTIONS:
Drug: Tofacitinib ointment — Patients with AA (with at least 2 patches of alopecia involving the scalp), AT or AU will be treated with tofacitinib ointment for a maximum of 6 months. During treatment, patients will be evaluated every 4 weeks and effectiveness of the medication will be measured by changes in hair growth.

SUMMARY:
The purpose of the study is to investigate the use of topical tofacitinib to promote hair regrowth in patients with alopecia areata, alopecia totalis, and alopecia universalis.

DETAILED DESCRIPTION:
This will be an open label clinical trial. We plan to treat 10 adults with AA (with at least 2 patches of alopecia involving the scalp), AT or AU with tofacitinib ointment for a maximum of 6 months. During treatment, patients will be evaluated every 4 weeks and effectiveness of the medication will be measured by changes in hair growth. Laboratory evaluation will be performed before and during treatment in order to monitor for adverse effects of the medication.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AA with at least 2 patches of alopecia involving the scalp, AT or AU
* Stable hair loss present for 6 months or longer
* No treatment for alopecia areata in the past 1 month
* No evidence of spontaneous hair regrowth

Exclusion Criteria:

* Patients have received treatment known to affect alopecia areata within 1 month of enrolling in the study
* Patients whose current episode of AT or AU is more than 5 years
* Patients with a history of malignancy (except history of successfully treated basal cell or squamous cell carcinoma of the skin)
* Patients known to be HIV or hepatitis B or C positive
* Patients with positive tuberculin skin test or positive QuantiFERON® TB test
* Patients with leukopenia or anemia
* Patients with renal or hepatic impairment
* Patients taking immunosuppressive medications, including but not limited to prednisone, methotrexate, mycophenolate mofetil, azathioprine, tacrolimus, cyclosporine, or TNF-α inhibitors
* Women who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-09; Primary Completion 2018-07 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett King, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bayart CB, DeNiro KL, Brichta L, Craiglow BG, Sidbury R. Topical Janus kinase inhibitors for the treatment of pediatric alopecia areata. J Am Acad Dermatol. 2017 Jul;77(1):167-170. doi: 10.1016/j.jaad.2017.03.024. No abstract available. PMID 28619556

RESULTS

PARTICIPANT FLOW:
Groups:
- Tofacitinib Ointment: Patients with alopecia areata (AA) (with at least 2 patches of alopecia involving the scalp), alopecia totalis (AT) or alopecia universalis (AU) will be treated with tofacitinib ointment for a maximum of 6 months. During treatment, patients will be evaluated every 4 weeks and effectiveness of the medication will be measured by changes in hair growth between baseline and the end of study.
  Tofacitinib ointment: Patients with AA (with at least 2 patches of alopecia involving the scalp), AT or AU will be treated with tofacitinib ointment for a maximum of 6 months. During treatment, patients will be evaluated every 4 weeks and effectiveness of the medication will be measured by changes in hair growth between baseline and end of study.
Period: Overall Study
Arm/Group | Tofacitinib Ointment
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tofacitinib Ointment
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
SALT score [Mean (Standard Deviation); unit: units on a scale] — SALT score range is from 0 (no hair loss) to 100 (100% hair loss)
  units on a scale | 77.7 (32.3)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Severity of Alopecia Tool (SALT) Score
Description: SALT score range is from 0 (no hair loss) to 100 (100% hair loss). A positive percent change from baseline corresponds to a reduction in SALT score, and in this study study will be measured between baseline and 6 months.
Time Frame: 6 Months
Measure: Mean (Full Range); unit: percent change
Arm/Group | Tofacitinib Ointment
Number analyzed (Participants) | 10
percent change | 10 [0 to 61]

2. Secondary Outcome: Treatment Response Assessed as the Number of Participants With Hair Regrowth
Description: Clinical photographs will be used to demonstrate presence or absence of hair regrowth. Presented is a count of people that did respond to treatment.
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Ointment
Number analyzed (Participants) | 10
Participants | 3

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Tofacitinib Ointment
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 7/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib Ointment (N=10)
Upper Respiratory Infection (Infections and infestations) | 4
Sinus Infection (Infections and infestations) | 1
Headache (General disorders) | 2
Folliculitis (Skin and subcutaneous tissue disorders) | 1
Scalp Skin Irritation (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT02812342/Prot_SAP_000.pdf